CLINICAL TRIAL: NCT00215566
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of Multiple Doses and Dose Levels of DDP733 in Patients With Irritable Bowel Syndrome With Constipation
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacodynamics of DDP733 for IBS-c
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dynogen Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DDP733-04-007
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2006-03

CONDITIONS: Irritable Bowel Syndrome With Constipation; Irritable Bowel Syndrome
Keywords: IBS; IBS-c
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — DDP733

INTERVENTIONS:
Drug: DDP733

SUMMARY:
This study will evaluate the safety, tolerability and pharmacodynamics of the investigational drug DDP733 in treating subjects with IBS-c. A placebo control will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a history of IBS-c for at least 3 months prior to randomization as assessed using ROME criteria
* Must have had endoscopic/radiologic bowel evaluation within the past 10 years
* Must comply with completing a daily diary and be able to comply with GI transit measurements, including swallowing capsules containing small x-ray visible markers
* Female subjects cannot be pregnant, post-partum for less than 1 year or breastfeeding

Exclusion Criteria:

* Serious underlying diseases, including psychiatric disorders
* Current history of conditions affecting bowel transit
* Recent history of biochemical or structural abnormalities of the gastrointestinal tract, gastrointestinal surgery, or gastrointestinal infection
* Clinically significant abnormal examination findings or laboratory tests
* Inability to stop taking certain medications, or a planned change in medications (including herbal remedies) which could interfere with study assessments
* Use of drugs and or ethanol which may interfere with compliance of study procedures or influence study outcome
* Presence of a medical condition which could interfere with the interpretation of study data
* Significant use of nicotine or caffeine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2005-09

PRIMARY OUTCOMES:
Evaluation of the effect of DDP733 on gastrointestinal transit

SECONDARY OUTCOMES:
Evaluation of the effect of DDP733 on patient reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: William Paterson, MD, Study Chair — Hotel Dieu Hospital
Locations (15):
- Canada (15):
  - Hys Medical Centre, Edmonton, Alberta
  - St Paul's Hospital, Vancouver, British Columbia
  - West Vancouver, British Columbia
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Surrey GI Clinic, Guelph, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario
  - St. Joseph's Healthcare, London, Ontario
  - Meadowlands Family Health Centre, Ottawa, Ontario
  - London Road Diagnostic Clinic, Sarnia, Ontario
  - Sarnia Institute of Clinical Research, Sarnia, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Toronto Digestive Disease Associates, Inc, Toronto, Ontario
  - Hopital St-Sacrement, Québec, Quebec